CLINICAL TRIAL: NCT02215447
Title: A Feasibility Study Of NAB-Paclitaxel In Combination With Carboplatin As First Line Treatment Of Gastrointestinal Neuroendocrine Carcinomas
Acronym: NABNEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barwon Health (Other Government)
Collaborators: Specialised Therapeutics Australia (Unknown); Deakin University (Other); Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCC 14.01
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Gastrointestinal Neuroendocrine Carcinomas
Keywords: NAB-paclitaxel; Gastrointestinal Neuroendocrine Carcinomas; phase II; carboplatin
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NAB-Paclitaxel with carboplatin (Experimental): NAB paclitaxel (100 mg/m2 IVI) every week (d1,8,15) in three weekly cycle. Carboplatin (AUC=5 IVI) (d1) in three weekly cycle. Study treatment will continue until progressive disease, unacceptable toxicity, or ceased by patient or clinician preference.
  Interventions: Drug: NAB paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: NAB paclitaxel — 100 mg/m2 i.v. every week (d1,8,15) in three weekly cycle Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Abraxane
Drug: Carboplatin

SUMMARY:
Gastrointestinal Neuroendocrine Tumours (NETs) are gaining increasing recognition as a highly prevalent disease, responsive to a number of therapies, some of which are proven in modern randomised controlled trials, but many of which still require high quality clinical trial evidence to confirm their effectiveness and guide their use in practice. This study is the first prospective trial to evaluate modern combination chemotherapy. The study will determine whether Carboplatin and Paclitaxel NAB is a suitable combination for comparison in a subsequent randomised controlled phase III international trial.

Given the paucity of randomized studies in NETs, there are no clear evidence based guidelines. Patients are treated according to guidelines established for small cell lung cancer, incorporating platinum (cisplatin or carboplatin) based doublet treatment with etoposide. Although these tumors are initially highly chemosensitive, the natural history of this disease is such that relapses occur early, which ultimately leads to a very poor prognosis. Almost all clinical trials investigating cytotoxic chemotherapy in NETs are small single arm studies and guidelines are derived from expert opinion and from extrapolating results from small cell lung cancer studies. Prospective clinical trials in this group of patients needs to be conducted to establish an evidence based standard of care and to improve the prognosis of this highly aggressive group of tumors.

Participants will receive albumin bound paclitaxel (ABRAXANE®) 100 mg/m2 administered as an intravenous infusion over 30 minutes on Days 1, 8, and 15 of each 21 day cycle. Carboplatin will be given at an Area Under the Curve (AUC) = 5 mg/min/mL on Day 1 only of each 21 day cycle administered over 30 mins, beginning immediately after the completion of albumin bound paclitaxel administration. Participants can continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.

DETAILED DESCRIPTION:
Gastrointestinal Neuroendocrine Tumours (NETs) are gaining increasing international recognition as a highly prevalent disease, responsive to a number of therapies, some of which are proven, but many of which still require high quality clinical trial evidence to confirm their effectiveness and guide their use in practice. This study is the first prospective trial to evaluate modern combination chemotherapy. Given the paucity of randomized studies in neuroendocrine carcinomas (NECs), there are no clear evidence based guidelines. Patients are treated according to guidelines established for small cell lung cancer. Although these tumors are initially highly chemosensitive, the natural history of this disease is such that relapses occur early, which ultimately leads to a very poor prognosis. Prospective clinical trials in this group of patients needs to be conducted to establish an evidence based standard of care and to improve prognosis. NETs are a heterogeneous group of malignancies originating from cells of the neural. They have a variable and often long natural history. They commonly arise from the gastrointestinal tract (58%), pancreas or lung (27%), and low grade NETs can be associated with symptoms resulting from the secretion of hormones or vasoactive peptides. NETs used to be thought of as rare but recently have been shown to be more common with rising incidence rates (3.3/100,000 in Australia 2000-2006). Prevalence (35/100, 000) is much higher than incidence resulting from five year survivorship of ~ 60% resulting in NETs being more prevalent than either gastric, pancreatic, oesophageal or hepatobiliary adenocarcinomas, or any 2 of these cancers combined. They can present multiple complex clinical challenges, thereby significantly contributing to cancer related morbidity and health costs in the Australian population. More recently, international interest groups such as the European Neuroendocrine Tumor Society have identified the need to establish a framework promoting opportunities for research and ensuring that the available evidence is incorporated into clinical practice guidelines.

Almost all clinical trials investigating cytotoxic chemotherapy in NECs are small single arm studies with guidelines derived from expert opinion and from extrapolating results from small cell lung cancer studies. Most guidelines recommend the combination of a platinum compound with etoposide. This combination is an established standard of care for small cell lung cancer, another tumour with neuroendocrine differentiation. However, the data are less clear for non-pulmonary neuroendocrine neoplasms (NENs) and NECs.

It is striking that almost all published NEC chemotherapy studies are non randomized and include relatively small numbers of patients often with heterogeneous pathology. Although there are no prospective studies with carboplatin and etoposide for NECs, it is remarkable that it is widely accepted as the standard chemotherapy for this disease.

A Phase 2 multi-center trial evaluating the efficacy of chemotherapy with paclitaxel, carboplatin and etoposide in advanced poorly differentiated NECs showed after 4 cycles of this combination treatment, patients who achieved an objective response or stable disease went on to have 24 weeks of weekly paclitaxel as maintenance treatment. Of the 78 patients treated, 15% had a complete response and the overall response rate was 53%. Five patients remained disease free from 18 to 66 months after therapy. The median survival was 14.5 months. However, the authors concluded that the 3 drug combination was moderately toxic and had no obvious efficacy advantage over the standard platinum/etoposide regimens.

This year (2013 ASCO) in an abstract a single European centre reported relative responses up to 50% in a retrospective series of NECs using 3 weekly paclitaxel, carboplatin and etoposide.

NAB paclitaxel is suggested to achieve a higher intracellular tumour paclitaxel concentration via the albumin mediated transendothelial transport system.

Participants will receive albumin-bound paclitaxel (ABRAXANE®) 100 mg/m2 administered as an intravenous infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle. Carboplatin will be given at an Area Under the Curve (AUC) = 5 mg/min/mL on Day 1 only of each 21-day cycle administered over 30 mins, beginning immediately after the completion of albumin-bound paclitaxel administration. Participants can continue treatment at the investigator's discretion until disease progression, development of an unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with unresectable neuroendocrine carcinoma
* Age ≥18 yrs
* Histologically proven neuroendocrine carcinoma (NEC) as defined by the WHO Classification of Tumours of the Digestive System, 4th Ed - including tumours mixed with other malignancies (i.e. MANEC or mixed NEC/SCC). The features of small versus large cell NEC carcinoma will need to be documented.
* Tumour sufficiently Fluorodeoxyglucose (FDG)-avid (SUVmax minimum 3.5) on the initial staging PET
* Patients with advanced and/ or metastatic disease
* Measurable disease as assessed by CT scan of the chest, abdomen and pelvis as per RECIST v 1.1, within 21 days prior to commencement of study treatment
* ECOG performance status 0-1
* Adequate haematological, renal and hepatic function (neutrophils ≥2 × 109/L, platelets ≥100 × 109/L, hemoglobin ≥100g/L, total bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase ≤2.5 × ULN, alkaline phosphatases ≤2.5 ULN, creatinine ≤ 1.5 ULN)
* Signed, written informed consent

Exclusion Criteria:

* NECs confirmed not to be from gastrointestinal primaries and NETs of lower grades (Ki67<20)
* Suspected pulmonary origin of the NET e.g., FDG-PET avid lung lesions in patients with NEC liver metastases.
* Known hypersensitivity to NAB paclitaxel
* External beam radiotherapy to solitary target lesions. Patients who have received local radiotherapy of non-target lesions for local symptom control within the last 4 weeks must have recovered from any adverse effects of radiotherapy prior to starting treatment.
* Prior intrahepatic 90Ymicrospheres such as SIR-Spheres
* Major surgery/surgical therapy for any cause within 1 month or surgical therapy of loco-regional metastases within the last 3 months prior to starting treatment
* Severe cardiovascular, hepatic, neurologic or renal comorbid conditions
* Previous cytotoxic chemotherapy, or targeted therapy, or biotherapy for NEC (prior Somatostatin analogs (SSAs) are allowed)
* History of hepatitis B or C
* Sensory/motor neuropathy ≥ to grade 2, as defined by NCI CTCAE 4.0
* Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a (double if required) barrier method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Response rate | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The objective tumour response rate (partial or complete response as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1) via CT until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Progression free survival | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The rate of progression free survival (PFS). (PFS defined from time of registration to disease progression as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1).
Overall survival | From date of registration until date of death from any cause, assessed up to 36 months
  Overall survival (OS) (death from any cause).
Rates of adverse events as defined by NCI- Common Terminology Criteria for Adverse Events (CTCAE) V4.0 | During study drug administration until 30 days after last study drug dose

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MD, Study Chair — Barwon Health
Locations (3):
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Barwon Health, Geelong, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria